CLINICAL TRIAL: NCT04910334
Title: Long-term Cognitive and Functional Status After COVID-19 Treatment at Danish ICUs
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-135-2020
Record Dates: First submitted 2021-02-04; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: covid-19; danish icu; long-term follow-up
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective observational cohort study of 6 and 12 months long-term outcome of Danish speaking patients with COVID-19.

DETAILED DESCRIPTION:
To describe frailty, cognitive function, functional status, fatigue, mortality and the quality of life 6 and 12 months after ICU admission of the COVID-19 patients enrolled in the Danish ICU COVID-19 database. Furthermore to investigate the association between ventilator days and Clinical Frailty Score (CFS) and the MiniMoCA, respectively at 6 and 12 months after ICU admission

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* enrolled in the 'Danish ICU COVID-19 database'

Exclusion Criteria:

* non danish speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is all Danish speaking COVID-19 patients, admitted and treated at one of the 29 Danish ICUs, and enrolled in the 'Danish ICU COVID-19 database' from March 10th and forward. Patients are 18 of age and above with a positive polymerase chain reaction (PCR) test for SARS-CoV-2 either prior to or during ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
The cognitive status at 6 and 12 months after ICU admission using the validated instrument MiniMoCA | at 6 and 12 months after ICU admission
  The cognitive status at 6 and 12 months after ICU admission using the validated instrument MiniMoCA. Score 0-15, score above 11 indicate normal cognitive function. Two time points to see if there is a change in the cognitive status over time.
The functional status at 6 and 12 months after ICU admission using the validated instrument CFS | at 6 and 12 months after ICU admission
  The functional status at 6 and 12 months after ICU admission using the validated instrument CFS (score 1-9) higher levels indicate more frailty. Two time points to see if there is a change in the frailty status over time.

SECONDARY OUTCOMES:
The association between ventilator days and CFS 6 and 12 months after ICU admission | at 6 and 12 months after ICU admission
  The association between ventilator days and CFS 6 and 12 months after ICU admission. Will be one analysis.
The association between ventilator days and MiniMoCA 6 and 12 months after ICU admission | at 6 and 12 months after ICU admission
  The association between ventilator days and MiniMoCA 6 and 12 months after ICU admission. Will be one analysis. But need to time points to see if there is a change.
Mortality 6 and 12 months after ICU admission | at 6 and 12 months after ICU admission
  Mortality 6 and 12 months after ICU admission. To see if there is a change i mortality at 6 and 12 months.
EQ-5D-5L score 6 and 12 months after ICU admission | at 6 and 12 months after ICU admission
  EQ-5D-5L score 6 and 12 months after ICU admission. Score 5-25. low score indicate better quality of life. Two time points to see if there is a change.
Barthel ADL score 6 and 12 months after ICU admission | at 6 and 12 months after ICU admission
  Barthel ADL score 6 and 12 months after ICU admission. Score 0-20, high score indicate high independence. Two time points to see if there is a change.
Lawton-Brody IADL score 6 and 12 months after ICU admission | at 6 and 12 months after ICU admission
  Lawton-Brody IADL score 6 and 12 months after ICU admission. score from 0-8 for female and 0-5 for male. High score indicate high independence. Two time points to see if there is a change.
FAS score 6 and 12 months after ICU admission | at 6 and 12 months after ICU admission
  FAS score 6 and 12 months after ICU admission. score from 10-50, high score indicate high level of fatigue. Two time points to see if there is a change.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Poulsen, MD, Study Director — Department of Anaesthesiology and Intensive Care
Locations (1):
- Department of Anaesthesiology, Køge, Denmark